CLINICAL TRIAL: NCT03690843
Title: The Development of Children With Developmental Coordination Disorder (DCD) Before the Age of Six: a Follow-up Study
Brief Title: Development of Children With DCD Before the Age of Six
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: B670201837290
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-12

CONDITIONS: Developmental Coordination Disorder
Keywords: motor development; toddler; prediction
MeSH Terms: conditions — Motor Skills Disorders | interventions — Body Mass Index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DCD Group: Children diagnosed with DCD or at-risk DCD at two or three years of age
  Interventions: Other: Test Battery
- Control Group: Typically developing children
  Interventions: Other: Test Battery

INTERVENTIONS:
Other: Test Battery — All toddlers (DCD children + TD children) included in the study will be tested at three points in time, that is at the age of 3y, 4y and 5y with an extensive test battery. Questionnaires will be filled in by parents and teachers. Children will be tested using different instruments.
  Other Names: Movement Assessment Battery for Children 2; Beery-VMI-6; Functional Strength Measurement; Child Behaviour Checklist; Little-DCD-Questionnaire; Teacher Report Form; DCD-Daily-Questionnaire; Vragenlijst motorische vaardigheden kleuters; Body mass Index; YC-PEM; Social Communication Questionnaire

SUMMARY:
The aim of this study is to map the early development of children with DCD and compare it to typically developing (TD) children.

At first we will investigate to what extent motor delay, reduced force, higher BMI, behavioral, ADL and participation problems occur in toddlerhood in DCD children and how this relates to TD children. We will also look into the evolution of these parameters in time (stability of development).

Secondly we will explore if the diagnosis of DCD can be predicted using a standardized test before the age of five.

DETAILED DESCRIPTION:
A longitudinal study design enables us to assess children at three different ages (3y, 4y and 5y).

Assessment scores (AIMS or/and BSID) before the age of three will be retrieved retrospectively in the clinical group.

ELIGIBILITY:
Inclusion Criteria DCD group:

1. The multidisciplinary team of the Center of Developmental Disabilities reports that the child has DCD or is at-risk for developing DCD and this at the age of 2 and/or 3 years.
2. At least one parent speaks Dutch to the child

Inclusion Criteria controlgroup:

1. The child is three years of age at the moment of the first testing
2. Little-DCD-Q score ≥ 55 at 3y
3. M-ABC-2 percentilescore ≥25 at 3y
4. No medical diagnoses possibly influencing the motor development (DCD, ADHD, ASS, CP,…)
5. No history of developmental motor stimulation (therapy) and/or support
6. Gestational age ≥37w
7. Birthweight ≥2500g
8. At least one parent speaks Dutch to the child

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children attending the Center of Developmental Disabilities Ghent.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2023-01-06 (Actual); Study Completion 2023-01-06 (Actual)

PRIMARY OUTCOMES:
Developmental Coordination Disorder | This will be assessed at the age of 5 years.
  Presence or absence of a diagnosis of DCD as defined by the DSM-V diagnostic criteria.

SECONDARY OUTCOMES:
Movement Assessment Battery For children 2 - Dutch Version | This will be assessed at the age of 3, 4 and 5 years.
  The M-ABC-2-NL is a motor assessment battery for children age 3 to 16y including three subtests (manual dexterity, ball skills and balance). The test battery was translated to Dutch and Dutch-Flemish norms are available.
Beery-Buktenica Developmental test of Visual-Motor Integration 6 | This will be assessed at the age of 3, 4 and 5 years.
  The Beery-VMI-6 measures the visual-motor integration skills and consists of three subtests (visual-motor integration, motor coordination and visual perception).
Child Behaviour CheckList | This will be assessed at the age of 3, 4 and 5 years.
  The CBCL consists of 120 items (3-pointscale) questioning the child's behavior. Two versions are available (teacher and parent) in two age-ranges (1.5y - 6y and 6y - 18y). The absence or presence of features of emotional disorder, anxiety disorder, AD(H)D, OCD, CD and somatic disorder are examined.
  Both versions (parent + teacher) within the age-range 1.5 - 6y will be used.
Functional Strength Measurement | This will be assessed at the age of 4 and 5 years.
  The FSM is a Dutch test assessing functional force in children 4 to 12y. The test consists of 8 items in two domains (upper extremity and lower extremity). Scores are presented either by limb (upper or lower limb) and/or by type of force (explosive power/endurance).
Young Children's Participation and Environment Measure | This will be assessed at the age of 3, 4 and 5 years.
  YC-PEM is a questionnaire for parents of children aged 0 to 6y. The test consists of 73 items on three participation scales (frequency, involvement and desire to change) and one environment scale (amount of support by environment) measured in three domains (home, kindergarden/school and community).
Little-DCD-Questionnaire | This will be assessed at the age of 3, 4 and 5 years.
  The L-DCD-Q-NL originates in Israel and was designed for children 3 to 4y. It is a revision of the DCD-Q for older children. The Flemish translation expanded the age category from 3 to 5y. The L-DCD-Q is a parental questionnaire scoring 15 activities using a 5-point-Likert scale.
Motor Skills Checklist (VMVK) | This will be assessed at the age of 3, 4 and 5 years.
  The VMVK is a Flemish teacher questionnaire consisting of 28 ADL-activities scored using a 4-point-scale. Norms are available for children age 3 to 5y.
DCD-Daily Questionnaire | This will be assessed at the age of 5 years.
  The DCD-Daily-Q is a Dutch parental questionnaire (5 - 8y) consisting of 23 ADL-activities (3-point scale) in three domains: how often the child participates (participation scale), how well the child performs (quality scale) and the time the child needs to learn new skills (learning scale).
Body Mass Index | This will be assessed at the age of 3, 4 and 5 years.
  Height and weight will be determined.
Social Communication Questionnaire | This will be assessed at the age of 5 years.
  SCQ is a parental screening questionnaire for autism in children aged 4 years or older. The questionnaire consists of 40 yes/no questions.
Teacher report form | This will be assessed at the age of 3, 4 and 5 years.
  The TRFconsists of 120 items (3-pointscale) questioning the child's behavior. Two versions are available (teacher and parent) in two age-ranges (1.5y - 6y and 6y - 18y). The absence or presence of features of emotional disorder, anxiety disorder, AD(H)D, OCD, CD and somatic disorder are examined.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Roubaix, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No